CLINICAL TRIAL: NCT01441960
Title: Optimal Control of Muscle Strength for Electroconvulsive Therapy: A Comparison of Succinylcholine Versus Rocuronium-induced Neuromuscular Blockade
Brief Title: Optimal Dose of Succinylcholine and Rocuronium for Electroconvulsive Therapy (ECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ala Nozari, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010P001154
Record Dates: First submitted 2011-09-20; First posted 2011-09-28 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Neuromuscular Blockade; ECT
Keywords: Succinylcholine; Rocuronium; ECT
MeSH Terms: interventions — Succinylcholine; Rocuronium

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Succinylcholine first, then Rocuronium (Experimental): Cross-over randomized controlled, assessor blinded clinical trial.
  Interventions: Drug: Succinylcholine; Drug: Rocuronium
- Rocuronium first, then succinylcholine (Experimental): Cross-over randomized controlled, assessor blinded clinical trial.
  Interventions: Drug: Succinylcholine; Drug: Rocuronium

INTERVENTIONS:
Drug: Succinylcholine — Succinylcholine will be given during the series of ECT treatments. The initial dose will be defined by the anesthesiologist in charge for clinical care. The Dixon's up and down method will be used in consecutive treatments. The investigators will switch to the second compound as soon as the patient has received one neuromuscular blocking agent dose that resulted in 'acceptable muscle relaxation', and another dose that resulted in 'unacceptable' conditions'.
  Other Names: Suxamethonium
Drug: Rocuronium — Rocuronium will be given during the series of ECT treatments. The initial dose will be defined by the anesthesiologist in charge for clinical care. The Dixon's up and down method will be used in consecutive treatments.

SUMMARY:
Electroconvulsive therapy (ECT) is the transcutaneous application of small electrical stimuli to the brain to produce generalized seizures for the treatment of selected psychiatric disorders such as severe depression. The aim of ECT is to induce a therapeutic tonic seizure where the person loses consciousness and has convulsions. Patients need general anesthesia and neuromuscular blockade to treat pain and avoid excessive tonic clonic motor contraction that might be associated with compression fractures. Neuromuscular blocking drugs (NMBD) are, therefore, administered after induction of general anesthesia to induce neuromuscular blockade. Despite the importance of NMBDs to provide optimal conditions for ECT treatment, the optimal NMBD dose to achieve acceptable neuromuscular blockade without excessive or untoward effects has not previously been identified in any study and in a prospective randomized fashion. The aim of this study is, therefore, to identify the optimal NMBD dose of two commonly used neuromuscular blocking agents (succinylcholine and rocuronium) in order to optimize the muscle strength modulation during ECT that facilitates ECT with the minimal side effects.

DETAILED DESCRIPTION:
Patients, who consent to participate in the study, will randomly receive either succinylcholine or rocuronium by utilizing the Dixon's up and down technique. For patient safety, the first dose of either agent will be defined by the anesthesiologist providing care, and subsequent doses will be incrementally increased or decreased by 10% based on the assessment of a psychiatrist blinded to dose, who uses a dichotomous scale to assess the quality of the ECT (acceptable and not acceptable). The investigators will switch to the second compound as soon as the patient has received one neuromuscular blocking agent dose that resulted in 'acceptable muscle relaxation', and another dose that resulted in 'unacceptable' conditions'.

Acceleromyography will be used for monitoring neuromuscular transmission. Following induction of general anesthesia, the TOF-Watch SX will be calibrated (mode 1, 50 mA), and train-of-four (TOF) stimulation (every 15 seconds) will be initiated and maintained until recovery of the T1 to 100% baseline. Non-invasive blood pressure, heart rate, peripheral oxygen saturation (SpO2), and time to recovery of spontaneous breathing will be measured during the procedure. In addition the investigators will measure stimulation parameters used to initiate ECT, as well as the duration of seizure as well as the entire procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18-80) scheduled for ECT treatment at the MGH

Exclusion Criteria:

* Contraindication to the use of neuromuscular blocking drugs (e.g. allergy, preexisting muscular disease, and history of malignant hyperthermia)
* Malnutrition, general weakness
* Neurological or neuromuscular disease, including paralysis
* Liver disease with liver function test 2x greater than upper normal limit
* Kidney disease with eGFR<60
* Electrolyte abnormalities with values outside of the normal range
* Pregnancy
* Cardiac disease or abnormal EKG
* Medications that affect seizure threshold or blood pressure response
* Unwilling to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Massachusetts General Hospital; Ala Nozari, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Cheam EW, Critchley LA, Chui PT, Yap JC, Ha VW. Low dose mivacurium is less effective than succinylcholine in electroconvulsive therapy. Can J Anaesth. 1999 Jan;46(1):49-51. doi: 10.1007/BF03012514. PMID 10078403
- [Background] Turkkal DC, Gokmen N, Yildiz A, Iyilikci L, Gokel E, Sagduyu K, Gunerli A. A cross-over, post-electroconvulsive therapy comparison of clinical recovery from rocuronium versus succinylcholine. J Clin Anesth. 2008 Dec;20(8):589-93. doi: 10.1016/j.jclinane.2008.06.006. PMID 19100931
- [Background] Wagner KJ, Mollenberg O, Rentrop M, Werner C, Kochs EF. Guide to anaesthetic selection for electroconvulsive therapy. CNS Drugs. 2005;19(9):745-58. doi: 10.2165/00023210-200519090-00002. PMID 16142990
- [Background] Eikermann M, Hunkemoller I, Peine L, Armbruster W, Stegen B, Husing J, Peters J. Optimal rocuronium dose for intubation during inhalation induction with sevoflurane in children. Br J Anaesth. 2002 Aug;89(2):277-81. doi: 10.1093/bja/aef177. PMID 12378667
- [Background] Miguel RV, Soto R, Dyches P. A double-blind, randomized comparison of low-dose rocuronium and atracurium in a desflurane anesthetic. J Clin Anesth. 2001 Aug;13(5):325-9. doi: 10.1016/s0952-8180(01)00282-3. PMID 11498311
- [Background] Reynolds LM, Lau M, Brown R, Luks A, Fisher DM. Intramuscular rocuronium in infants and children. Dose-ranging and tracheal intubating conditions. Anesthesiology. 1996 Aug;85(2):231-9. doi: 10.1097/00000542-199608000-00002. PMID 8712436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 hospitalized patients aged 24-80 admitted for a series of ECT treatments at a frequency of 3/week were enrolled. 14 were excluded (1 received rocuronium in error, 1 received succinylcholine in error, 1 withdrew consent, 2 did not complete series of ECT, and in 9 twitch monitoring problems resulted in non-captured or disqualified data.
Pre-assignment Details: Patients were randomized to either succinylcholine or rocuronium during their first ECT. During each subsequent ECT ( 2 days apart) patients received a 10% higher (if insufficient paralysis) or lower dose (if sufficient or excessive paralysis) until the minimum effective dose was identified. Then the second NMBA was tested for subsequent ECTs.
Groups:
- Succinylcholine First, Then Rocuronium: After induction of anesthesia Succinylcholine (Quelicin®, Hospira Inc., Lake Forest, IL) 0.8 (2.67 × ED95) mg/kg was administered intravenously over 5 sec via an intravenous catheter in the arm contralateral to the side of neuromuscular transmission monitoring, which was then flushed with a 10 ml bolus of normal saline.
  By identifying the optimal (minimal effective) dose of succinylcholine, Rocuronium bromide (Zemuron®, Oganon USA Inc) 0.4 mg/kg (1.33 × ED95) was administered intravenously over 5 sec via an intravenous catheter in the arm contralateral to the side of neuromuscular transmission monitoring, which was then flushed with a 10 ml bolus of normal saline. After the ECT treatment and when appropriate, as determined by the practicing anesthesiologist, the induced neuromuscular blockade was reversed with neostigmine 50 microgram/kg, administered with glycopyrrolate 10 microgram/kg.
- Rocuronium First , Then Succinylcholine: After induction of anesthesia Rocuronium (Zemuron®, Oganon USA Inc) 0.4 mg/kg (1.33 × ED95) mg/kg was administered intravenously over 5 sec via an intravenous catheter in the arm contralateral to the side of neuromuscular transmission monitoring, which was then flushed with a 10 ml bolus of normal saline. After the ECT treatment and when appropriate, as determined by the practicing anesthesiologist, the rocuronium-induced neuromuscular blockade was reversed with neostigmine 50 microgram/kg, administered with glycopyrrolate 10 microgram/kg.
  By identifying the optimal (minimal effective) dose of rocuronium, in the subsequent treatment of the subject, Succinylcholine (Quelicin®, Hospira Inc., Lake Forest, IL) 0.8 (2.67 × ED95) mg/kg was administered intravenously over 5 sec via an intravenous catheter in the arm contralateral to the side of neuromuscular transmission monitoring, which was then flushed with a 10 ml bolus of normal saline.
Period: First Neuromuscular Blocking Agent:
Arm/Group | Succinylcholine First, Then Rocuronium | Rocuronium First , Then Succinylcholine
Started | 26 | 19
Completed | 18 | 13
Not Completed | 8 | 6
Not completed — Technical error or incomplete ECT series | 6 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Neuromuscular Blocking Agent
Arm/Group | Succinylcholine First, Then Rocuronium | Rocuronium First , Then Succinylcholine
Started | 18 | 13
Completed | 18 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Succinylcholine and Rocuronium: All study participants
Arm/Group | Succinylcholine and Rocuronium
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Optimal Dose of Neuromuscular Blocking Agent During ECT
Description: The optimal dose of muscle neuromuscular blocking is defined as the lowest dose of either compound that predicts 'acceptable' control of muscle strength during ECT. Assessment of the primary end point is based on a dichotomous scale 'acceptable' and 'not acceptable' control of muscle strength during ECT, and the two assessors will be blinded to the dose of neuromuscular blocking agent. The optimal dose was identified for each subject, and results were reported as the average of all lowest doses collected in the study.
Time Frame: Up to six weeks following inclusion
Measure: Mean (95% Confidence Interval); unit: mg.kg-1
Groups:
- NMBA: Sux: Cross-over randomized controlled, assessor blinded clinical trial.
  Succinylcholine: Succinylcholine will be given during the series of ECT treatments. The initial dose will be defined by the anesthesiologist in charge for clinical care. The Dixon's up and down method will be used in consecutive treatments. The investigators will switch to the second compound as soon as the patient has received one neuromuscular blocking agent dose that resulted in 'acceptable muscle relaxation', and another dose that resulted in 'unacceptable' conditions'.
- NMBA- Rocuronium: Cross-over randomized controlled, assessor blinded clinical trial. Rocuronium: Rocuronium will be given during the series of ECT treatments. The initial dose will be defined by the anesthesiologist in charge for clinical care. The Dixon's up and down method will be used in consecutive treatments.
Arm/Group | NMBA: Sux | NMBA- Rocuronium
Number analyzed (Participants) | 31 | 31
mg.kg-1 | 0.85 [0.77 to 0.94] | 0.41 [0.36 to 0.46]

2. Secondary Outcome: Compound Specific Differences in Time to Recovery From Neuromuscular Blockade
Description: The investigators defined the compound specific differences in time to recovery from neuromuscular blockade - i.e., recovery of spontaneous breathing and recovery of the twitch height to baseline.
Time Frame: Up to six weeks following inclusion
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Succinylchline; Rocuronium: Time to recovery after single bolus administered at the beginning of ECT therapy
Arm/Group | Succinylchline | Rocuronium
Number analyzed (Participants) | 31 | 31
minutes | 9.7 (3.5) | 19.5 (5.7)

3. Secondary Outcome: Differences in Seizure Duration Between Compounds
Description: Observational reports suggest that differences in seizure duration might exist depending on the neuromuscular blocking agents used to accomplish muscle strength control during ECT.
Time Frame: Up to six weeks following inclusion
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Succinylcholine: Duration of induced seizure after standard ECT
- Rocuronium: Duration of induced seizure
Arm/Group | Succinylcholine | Rocuronium
Number analyzed (Participants) | 31 | 31
Seconds | 27 (14) | 31 (11)

ADVERSE EVENTS:
Groups:
- NMBA: Succinylcholine; NMBA: Rocuronium: No adverse events occurred during the study
Arm/Group | NMBA: Succinylcholine | NMBA: Rocuronium
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No